CLINICAL TRIAL: NCT03497364
Title: Improving Combined Spinal-epidural Anesthesia for Decreasing Hypotension in Pregnant Women Without Prophylactical Prehydration and Vasopressors
Brief Title: Combined Spinal-epidural Anesthesia for Cesarean Section Without Prophylactical Prehydration and Vasopressors
Acronym: CSEAFCSWPPAV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: SZY-00251
Record Dates: First submitted 2018-03-22; First posted 2018-04-13 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Cesarean Section; Anesthesia, Spinal
Keywords: Cesarean Section; Hypotension; Combined spinal-epidural anesthesia
MeSH Terms: conditions — Hypotension | interventions — Bupivacaine; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bupivacaine group (Experimental): Pregnant women received combined spinal-epidural anesthesia by injecting bupivacaine. The dose of bupivacaine depended on height of subjects.
  Interventions: Drug: bupivacaine
- Ropivacaine group (Experimental): Pregnant women received combined spinal-epidural anesthesia by injecting ropivacaine. The dose of ropivacaine depended on height of subjects).
  Interventions: Drug: ropivacaine
- Control group (No Intervention): Pregnant women received combined spinal-epidural anesthesia by injecting bupivacaine. 2ml bupivacaine (0.75% bupivacaine (2 ml) + cerebrospinal fluid (1 ml)) was injection for all subjects.

INTERVENTIONS:
Drug: bupivacaine — 0.5 % bupivacaine (0.75% bupivacaine (2 ml) + cerebrospinal fluid (1 ml)) was injection according to the height of subjects (1.7 ml for 173~174cm, 1.65 ml for 170~172cm, 1.6 ml for 168~169cm, 1.55 ml for 165~167cm, 1.5 ml for 163~164cm, 1.45 ml for 160~162cm, 1.4 ml for 158~159cm, 1.35 ml for 155~157cm, 1.3 ml for 153~154cm, 1.25 ml for 150~152cm, 1.2 ml for 148~149cm)，1.15 ml for 145~147cm).
  Arms: Bupivacaine group
Drug: ropivacaine — 0.5 % ropivacaine (1% ropivacaine (1.5 ml) + cerebrospinal fluid (1.5 ml)) was injection according to the height of subjects (2.300 ml for 173~174cm, 2.225 ml for 170~172cm, 2.15 0ml for 168~169cm, 2.075 ml for 165~167cm, 2.000 ml for 163~164cm, 1.925 ml for 160~162cm, 1.850 ml for 158~159cm, 1.775 ml for 155~157cm, 1.700 ml for 153~154cm, 1.625 ml for 150~152cm, 1.55 0ml for 148~149cm, 1.475 ml for 145~147cm)
  Arms: Ropivacaine group

SUMMARY:
Hypotension is a common complication in pregnant women after spinal anesthesia and related with the dose of local anesthetic. Injecting small dose local anesthetic into subarachnoid space can decrease the incidence of hypotension, but increase the risk of incomplete analgesia and muscle relaxation. The investigators hypothesize there is an optimal dose of bupivacaine and ropivacaine for subarachnoid injection in pregnant women, which can cause enough anesthesia and obviously decrease the incidence of hypotension without prophylactical prehydration and vasopressors. To verify this hypothesis, full-term pregnant women who were scheduled for elective cesarean section were recruited.Combined spinal-epidural anesthesia was performed for pregnant women after written informed consents. The dose of bupivacaine or ropivacaine is small and depends on height of pregnant women. The blood pressure, heart rate, respiratory rate, SpO2 and fetal heart rate were recorded and the blood flow volume of uterine artery was monitored The sensory and motor block were evaluated. After delivery, umbilical blood samples were taken for blood gas analysis. APGAR scores and neurological behavior of infant were evaluated and recorded. In the intraoperative period, side-effects and requirement for sedation, epidural injection or general anesthesia were noted. The quality of anaesthesia (judged by the anaesthetist), the quality of muscle relaxation (judged by the surgeon) and the degree of intraoperative comfort (judged by the patient) were recorded as excellent, good, fair or poor.

DETAILED DESCRIPTION:
1. General: This was a single-centre randomized controlled trial performed at ShenZhen People's Hospital of Jinan University. Study protocol was approval was by the Ethics Committee of ShenZhen People's Hospital of Jinan University, ShenZhen, China (Permit No. SZY-00251, Chairperson Prof. Xiaofang Yu) on 8 February 2017. Pregnant women who were scheduled for cesarean section were recruited. Written informed consents were obtained from all patients. Women with cardiovascular disease, fetal abnormalities, placental abruption, placenta previa, placental abnormalities, sidewall placenta, abnormal fetal heart rate and spinal anesthesia contraindications were excluded from the study.
2. Sample Size Calculation: SBP < 90 mmHg or 70% of the baseline value is defined as hypotension; in the study by Langesaeter et al in Anesthesiology magazine, the incidence of hypotension was 20% with prophylactic phenylephrine, and we considered a ≤ 8% difference in the incidence of hypotension to be of clinical significance. Assuming a type I error protection of 0.05 and a power of 0.80, the sample size for a non-inferiority test (margin Δ=0.08) was estimated using the normal approximation to the binomial distribution. Therefore, each group requires 310 subjects.
3. Anesthesia: Women were randomly divided into three groups, Bupivacaine group, Ropivacaine group and Control group. After entering the operation room, patients were placed supine with left lateral tilt and blood pressure was measured three times at 1-min intervals. The arithmetic average of the three measured values was regarded as the basal pressure of pregnant women. Next, electrocardiogram and pulse oximetry were also monitored. Supplementary oxygen was given through a facemask. Venipuncture was performed in the forearm vein. In Bupivacaine and Ropivacaine group, 500 ml Ringer's lactate was slow given for subjects before anesthesia without prehydration. In Control group, 1000 ml hydroxyethylstarch (6%) was first infused for subjects in the ward, after that 500 ml Ringer's lactate was slow given for subjects before anesthesia.

   Then, with the subjects in left lateral position, combined spinal-epidural anesthesia was performed as follows: skin was infiltrated by lidocaine at the L3-4 or L4-5 interspace; epidural puncture needle was slowly perpendicularly advanced until the tip passed through the ligamentum flavum and reached to epidural space, which was verified with the loss-of-resistance; then intrathecal injection was carried out by spinal needle of 25G, and the epidural catheter was inserted 4-6 cm. Subjects were then immediately recovered in supine with left lateral tilt. In Bupivacaine group, 0.5 % bupivacaine (0.75% bupivacaine (2 ml) + cerebrospinal fluid (1 ml)) was injection. The dose of bupivacaine depended on height of subjects (1.7 ml for 173~174cm, 1.65 ml for 170~172cm, 1.6 ml for 168~169cm, 1.55 ml for 165~167cm, 1.5 ml for 163~164cm, 1.45 ml for 160~162cm, 1.4 ml for 158~159cm, 1.35 ml for 155~157cm, 1.3 ml for 153~154cm, 1.25 ml for 150~152cm, 1.2 ml for 148~149cm)，1.15 ml for 145~147cm). In Ropivacaine group, 0.5 % ropivacaine (1% ropivacaine (1.5 ml) + cerebrospinal fluid (1.5 ml)) was injection. The dose of ropivacaine depended on height of subjects (2.3 ml for 173~174cm, 2.2 ml for 170~172cm, 2.1ml for 168~169cm, 2.0 ml for 165~167cm, 1.9 ml for 163~164cm, 1.8 ml for 160~162cm, 1.7 ml for 158~159cm, 1.6 ml for 155~157cm, 1.5 ml for 153~154cm, 1.4 ml for 150~152cm, 1.3 ml for 148~149cm, 1.2 ml for 145~147cm). In Control group, 2ml bupivacaine (0.75% bupivacaine (2 ml) + cerebrospinal fluid (1 ml)) was injection for all subjects. Immediately after intrathecal injection, in control group, phenylephrine was introduced by continuous infusion pumps programmed for an infusion rate of 0.25 ug.kg-1.min-1 to maintain systolic blood pressure at ≥ 90 mmHg or 70% -100 % of baseline value. In Bupivacaine and Ropivacaine group, no prophylactic phenylephrine was introduced For all subjects, when systolic blood pressure was less than 90 mmHg or 70% of baseline value. 100 ug phenylephrine was given and repeated every 1 min until the systolic blood pressure returned to normal. When heart rate was less than 60 beat/min. 0.5-1mg atropine was given to maintain normal heart rate. Nausea and vomiting were treated with metoclopramide 10 mg i.v. Sensory block level after intrathecal injection was assessed with a 20G hypodermic needle (no sensation to pinprick). When the maximum sensory block height was lower than T8, epidural injection of 2% lidocaine (3ml/5min, total volume was less than 15 ml) was given or anesthetic technique was changed into general anesthesia.
4. Data acquisition: After intrathecal injection, the blood pressure, heart rate, respiratory rate, SpO2 and fetal heart rate were recorded every 1 min until fetal delivery and then were recorded every 3 min until the end of surgery. The blood flow volume of uterine artery was monitored by ultrasound.

   The level of sensory block, defined as the loss of pin-prick sensation (20G hypodermic needle) at midclavicular level, was measured every 1 min until it reached the T8 dermatome level and then every 10 min during surgery. The following variables were recorded: time to initial onset of analgesia, time for sensory block to reach the T8 dermatome level, time for sensory block to reach maximum dermatome level, time to two-segment regression of analgesic level, and regression of analgesic level to the S2 dermatome. Anesthesia was considered adequate for surgery if pain sensation was lost at the T8 level.

   Motor block was assessed every 1 min using the Bromage scale (0 = no motor block, 3 = complete motor block of lower limbs) until complete motor block and then every 30 min until the return of normal motor function. The times to complete motor block and complete recovery were recorded. The motor block score when the sensory block level reached T8 was also recorded.

   The time from anesthesia initiation to delivery, time from skin incision to delivery and time from uterus incision to delivery were recorded. The total dose of phenylephrine and total volume of fluid before delivery were recorded. After delivery, umbilical blood samples were taken for blood gas analysis. APGAR scores at 1 and 5 min were evaluated and recorded. In the intraoperative period, side-effects and requirement for sedation, epidural injection or general anesthesia were noted.

   Neurologic assessment (muscle force, muscle tone, sucking reflex, rooting reflex, moro reflex and grasp reflex) of the infant was carried out at 2h,4h,8h, 1d,2d,3d,4d and 7d after delivery. The quality of anaesthesia (judged by the anaesthetist), the quality of muscle relaxation (judged by the surgeon) and the degree of intraoperative comfort (judged by the patient) were recorded as excellent, good, fair or poor.
5. Statistical Analysis: Statistical analysis was performed using SPSS 13.0 software package. All metering data were recorded as mean ± standard deviation and Independent-Samples T test or One-way ANOVA was used to compare the metering data. Chi-square test was used to compare the enumeration data. p<0.05 indicates that the differences have statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who were scheduled for cesarean section.

Exclusion Criteria:

* Women with cardiovascular disease, fetal abnormalities, placental abruption, placenta previa, placental abnormalities, sidewall placenta, abnormal fetal heart rate and spinal anesthesia contraindications.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 930 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of hypotension after anesthesia | delivery
  Hypotension after anesthesia expressed in number of patients with one or more episodes of hypotension (Systolic blood pressure < 90 mmHg or 70% of baseline value) up to fetal delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Zhongjun Zhang, master, Study Director — ShenZhen People's Hospital of Jinan University
Locations (1):
- ShenZhen People's Hospital of Jinan University, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang J, Wen G, Huang Q, Huang B. Anesthesia characteristic of an algorithm of bupivacaine dose based on height in caesarean section under spinal anesthesia: a retrospective cohort study. BMC Anesthesiol. 2023 May 2;23(1):146. doi: 10.1186/s12871-023-02113-0. PMID 37131191
- [Derived] Huang Q, Wen G, Hai C, Zheng Z, Li Y, Huang Z, Huang B. A Height-Based Dosing Algorithm of Bupivacaine in Spinal Anesthesia for Decreasing Maternal Hypotension in Cesarean Section Without Prophylactic Fluid Preloading and Vasopressors: A Randomized-Controlled Non-Inferiority Trial. Front Med (Lausanne). 2022 Jun 10;9:858115. doi: 10.3389/fmed.2022.858115. eCollection 2022. PMID 35755061
- [Derived] Huang B, Huang Q, Hai C, Zheng Z, Li Y, Zhang Z. Height-based dosing algorithm of bupivacaine in spinal anaesthesia for decreasing maternal hypotension in caesarean section without prophylactic fluid preloading and vasopressors: study protocol for a randomised controlled non-inferiority trial. BMJ Open. 2019 May 16;9(5):e024912. doi: 10.1136/bmjopen-2018-024912. PMID 31101694